CLINICAL TRIAL: NCT02474979
Title: Reduced Pressure for Less Pressure Ulcers. Effect of the CBPM-system in a Swedish University Hospital
Brief Title: Reduced Pressure for Less Pressure Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Wellsense USA Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EPN2014/529
Record Dates: First submitted 2015-05-27; First posted 2015-06-18 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Pressure Ulcer
Keywords: Pressure ulcer; Prevention; Pressure mapping
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBPM-system (Experimental): CBPM-system (Continuous Bedside Pressure Mapping System): the bed is equipped with a pressure sensing mat including thousands of sensors. It is connected with a monitor that continuously registers the pressure between the body and the bed surface (interface pressure). The pressure is indicated by colors, where warmer colors indicate higher pressure. The CBPM-system will be used in addition to standard pressure ulcer prevention (PU reducing mattress, floating heels, repositioning).
  Interventions: Device: CBPM-system
- Control (Experimental): Standard pressure ulcer prevention (PU reducing mattress, floating heels, repositioning).
  Interventions: Other: Control

INTERVENTIONS:
Device: CBPM-system — The bed is equipped with a pressure sensing mat including thousands of sensors. It is connected with a monitor that continuously registers the pressure between the body and the bed surface (interface pressure). The pressure is indicated by colors, where warmer colors indicate higher pressure.
  Arms: CBPM-system
Other: Control
  Arms: Control

SUMMARY:
Pressure ulcers (PU) cause pain and discomfort to affected patients, as well as considerable costs for society. The present study will evaluate the effect of the Continuous Bedside Pressure Mapping (CBPM)- system on PU prevalence and incidence. A RCT including 180 patients will be conducted in a geriatric setting in a Swedish University hospital

DETAILED DESCRIPTION:
Background The first national PU prevalence study in Sweden conducted in 2011 showed a prevalence of 16.6% (n=16 466) in hospital settings. High age and reduced mobility/activity are main risk factors. International evidence-based guidelines for prevention of PU are available. Pressure relief (e.g repositioning, mattresses, chair cushions, heel cushions) is the main stay of preventive measures. Recent research shows that PU prevention is not a high priority. For example, the corner stone of prevention, repositioning, is not conducted for risk patients.

Aim To evaluate the effect of the CBPM-system on the prevalence and incidence of PU in hospital setting

Method Design: A randomised controlled trial will be conducted Sample: All patients admitted to the geriatric unit. Intervention: The CBPM-system will be used from admittance to discharge (not more than 14 days). Standard PU prevention (PU reducing mattress, floating heels, repositioning) Control group: Standard PU prevention (PU reducing mattress, floating heels, repositioning) Randomisation: Sealed envelopes will be used. Procedure: Two study nurses are responsible for inclusion of patients and data collection on day 1,3,7 and discharge. A photo will be taken of any PU. A PU expert will assess the photos after completed data collection (PU category 1-4). She will be blinded to group allocation.

Power calculation: The primary outcome of interest is the PU prevalence. Previous point prevalence studies in this geriatric unit shows a prevalence of 45%. The investigators goal is that the CBPM-system results in 20% decrease in the PU prevalence. In order to have 80% power to detect such a decrease with a two-sided two-sample proportions test at the 5% level, 89 patients per treatment group is needed. Intention-to-treat principals will be used.

Discussion The prevalence of PU, as well as prevention to risk patients are quality indicators in health care. National studies reveal an urgent need for quality improvement, New nursing methods and equipment must be systematically and scientifically evaluated.The results of this study will be valuable for nursing education and in international and national patient safety work to prevent PU. The results will also be valuable for other health professionals (physicians, physical and occupational therapists).

ELIGIBILITY:
Inclusion Criteria:

* Admitted to geriatric unit 30A during Sunday after 4 pm to Friday until 4 pm

Exclusion Criteria:

* Expected to be discharged before data collection in day 3

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2015-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
PU prevalence (Category 1-4) - change from baseline | admission to discharge or last assessment at 14 days
  The most severe PU for each patient is included in the calculation

SECONDARY OUTCOMES:
Number of PU per category and patient | admission to discharge or last assessment at 14 days
  Category 1-4
Number of preventive interventions | admission to discharge or last assessment at 14 days
  pressure reducing mattress, heel cushions, repositioning, repositioning aid, preventive dressing
Patient´s experience of comfort in bed | admission to discharge or last assessment at 14 days
  Visual Analog Scale 1-10
Peak pressure | admission to discharge or last assessment at 14 days
  mmHg (mean)

CONTACTS AND LOCATIONS:
Overall Officials: Lena Gunningberg, Professor, Principal Investigator — Uppsala University, Uppsala, Sweden
Locations (1):
- Akademiska sjukhuset, Uppsala, Uppland, Sweden